CLINICAL TRIAL: NCT06661707
Title: Comparative Study Between Ultrasound Guided Quadratus Lumborum Versus Ilioingunial/ Iliohypogastric Nerves Block as Post-operative Analgesia for Patients Undergoing Inguinal Hernia Repair Surgeries
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, RAMY AHMED, Assistant Professor of Anesthesia, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Ain Shams university S2
Record Dates: First submitted 2024-10-25; First posted 2024-10-28 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2024-10

CONDITIONS: Post Operative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Quadratus Lumborum block (QL) group (Active Comparator)
  Interventions: Procedure: Sonar guided Quadratus Lumborum block
- Ilioinguinal/Iliohypogastric block (ILI/IHG) group (Active Comparator)
  Interventions: Procedure: Sonar guided Ilioinguinal/Iliohypogastric block

INTERVENTIONS:
Procedure: Sonar guided Quadratus Lumborum block — The probe will be tilted down the lateral abdomen to identify a bright hyperechoic line that represents the middle layer of the thoracolumbar fascia. The needle will be inserted in plane from anterolateral to posteromedial. The needle tip will be placed between the thoracolumbar fascia and the QL muscle, and after negative aspiration, the correct position of the needle will be proved by injection of 5 mL of normal saline to confirm the space with a hypoechoic image and hydrodissection. An injection of (0.2 mL/kg of 0.25% bupivacaine per side) will be applied without exceeding the toxic dose 3 mg/kg
  Arms: Quadratus Lumborum block (QL) group
Procedure: Sonar guided Ilioinguinal/Iliohypogastric block — The ultrasound linear probe will be placed over the anterior superior iliac spine with the superior margin of the transducer pointed directly in an oblique plane toward the umbilicus. The iliohypogastric nerve will be seen medial to the ilioinguinal nerve. The overlying skin will be prepared with antiseptic solution and 21 gauge 120mm Locoplex Sono Tap cannula will be advanced using an in-plane approach from a point just below the inferior border of the transducer toward the ilioinguinal nerve as it lies within the facial plane between the internal abdominal oblique and transverse abdominis muscles.
  After negative aspiration, (0.2 mL/kg of 0.25% bupivacaine per side) will be injected without exceeding the toxic dose of 3 mg/kg
  Arms: Ilioinguinal/Iliohypogastric block (ILI/IHG) group

SUMMARY:
Postoperative pain management is becoming an integral part of anesthesia care. Various techniques of pain relief have been designed. We have designed the study for comparison between ultrasound guided quadratus lumborum (QL) block versus Ultrasound-guided ilioinguinal and iliohypogastric nerves (ILI+IHG) block as regard postoperative pain block and opioid consumption in patients undergoing inguinal hernia repair under general anesthesia.

DETAILED DESCRIPTION:
In the anesthesia clinic, an informed written consent will be taken from every patient one day before the surgery. Explanation of the visual analogue score (VAS) will be performed. History, clinical examination and routine investigations including; complete blood count (CBC), fasting blood sugar (FBS), liver function test (LFT), kidney function test (KFT), electrocardiogram (ECG), prothrombin time (PT) and activated partial thromboplastin time (aPTT) will be performed to all patients.

In the induction room, an intravenous (IV) 20 gauge cannula will be inserted and premedication will be limited to intravenous (IV) midazolam (0.03 mg/kg).

* Intra-operative setting:
* General anesthesia technique:

The patient will be fasting for at least 8 hours preoperatively. A standardized general anesthesia protocol will be used for all patients. General anesthesia will be induced with propofol (1.5-2 mg /kg) and fentanyl (1 µg /kg) with neuromuscular block Atracurium (0.5mg/kg at induction then 0.1mg/kg as maintenance dose. The patient's airway will be maintained using an endotracheal tube. Maintenance of anesthesia will be commenced using isoflurane (1.2%) in a 50% mixture of oxygen in air.

Ventilator Settings: the ventilation will be achieved with a volume-controlled mode ventilation, respiratory rate adjusted according to EtCO2 to range between 30-35 mmHg, a tidal volume of 6-8 ml/kg and mixture of gases in proportion 50% oxygen and 50% air, with PEEP 5 cm H2O using a closed circle system with a total fresh gas flow rate of 3L/min.

All patients will receive Ondansetron 8mg IV as antiemetic prophylaxis. Fentanyl (0.5 µg /kg) will be given for intraoperative rescue analgesia in case of tachycardia (heart rate more than 90 bpm or more than 20% of the base line of the patient) or hypertension (blood pressure more than 139/89mmHg or more than 20% of the base line of the patient) due to intraoperative pain after exclusion of other causes of tachycardia and increased blood pressure. 1 gm paracetamol will be given 30 minutes before skin closure.

Study procedures (The intervention): (The procedure will be done by the most experienced member of the research team) The procedure will be done in the operating rooms (OR) under complete aseptic technique by the most experienced member of the research team. Patients will be randomly allocated by computer generated randomization to one of the two groups according to the used block into

Group A; Quadratus Lumborum block (QL) group Group B; Ilioinguinal/Iliohypogastric block (ILI/IHG) group

Preparations that will be used for each patient are:

* Sterile towels, sponges, 4-inch gauze packs and povidone iodine 5% for sterilization, sterile gloves and 21gauge 120mm Locoplex Sono Tap cannula (Locoplex@ VYGON, France).
* The study drugs (commercially available forms) that will be used are:
* A 20 ml vial of 0.5% (bupivacaine hydrochloride).
* A 50ml vial of 2% (Lidocaine hydrochloride).

Group A; Quadratus Lumborum block (QL) group (22 patients) :

The patient will be positioned supine with lateral tilt to perform the block, and the transducer will be placed at the level of the anterior superior iliac spine and will be moved cranially until the three abdominal wall muscles will be clearly identified. The external oblique muscle will be followed postero-laterally until its posterior border will be visualized (hook sign), leaving underneath the internal oblique muscle, like a roof over the QL muscle. The probe will be tilted down to identify a bright hyperechoic line that represents the middle layer of the thoracolumbar fascia. The needle will be inserted in plane from anterolateral to posteromedial. The needle tip will be placed between the thoracolumbar fascia and the QL muscle, and after negative aspiration, the correct position of the needle will be proved by injection of 5 mL of normal saline to confirm the space with a hypoechoic image and hydrodissection. An injection of (0.2 mL/kg of 0.25% bupivacaine per side) will be applied without exceeding the toxic dose 3 mg/kg.

Group B; Ilioinguinal/Iliohypogastric block (ILI/IHG) group (22 patients):

The ultrasound linear probe will be placed over the anterior superior iliac spine with the superior margin of the transducer pointed directly in an oblique plane toward the umbilicus. The iliohypogastric nerve will be seen medial to the ilioinguinal nerve. The overlying skin will be prepared with antiseptic solution and 21 gauge 120mm Locoplex Sono Tap cannula will be advanced using an in-plane approach from a point just below the inferior border of the transducer toward the ilioinguinal nerve as it lies within the facial plane between the internal abdominal oblique and transverse abdominis muscles.

After negative aspiration, (0.2 mL/kg of 0.25% bupivacaine per side) will be injected without exceeding the toxic dose of 3 mg/kg.

o Postoperative settings: At the end of the procedure, the residual neuromuscular block will be reversed with injection of neostigmine (0.05 mg/kg) with atropine (0.01 mg/kg intravenous). Endotracheal tube extubation will be done after oral and endotracheal suction, then the patient will be transferred to postoperative anesthesia care unit (PACU).

At the post-anesthesia care unit (PACU) all patients will receive standard protocol of intravenous paracetamol 1 gm every 6 hours for the following 24 hours, and rescue dose of IV pethidine 50 mg if VAS score is ≥3.

If VAS score is ≥3 after 2 hours another dose of pethidine 25mg IM will be given and repeated if VAS score remains ≥3 every 2 hours for 24 hours postoperatively.

In the surgical ward vital signs (heart rate and blood pressure) as well as pain intensity will be assessed every 2 hours for 24 hours postoperatively.

o If local anaesthetic toxicity occurred, cardiovascular and respiratory support and 20% intralipid bolus of 100 ml over 2-3 min will be given.

ELIGIBILITY:
Inclusion Criteria:

* Physical Status: ASA (American society of Anesthesiologists) I - II patients.
* undergoing inguinal hernia repair

Exclusion Criteria:

* Contraindications to QL block & ILI+IHG nerve block such as; (Infection at site of injection, allergy to local anesthetic drugs.)
* Refusal of procedure or participation in the study by patients.
* Psychiatric illness or uncooperative patient.
* Coagulopathy, use of anticoagulants or antiplatelet therapy.
* Chronic analgesic users, drug addicts and alcoholic patients.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Estimated)
Dates: Start 2024-10-30 (Estimated); Primary Completion 2025-05-30 (Estimated); Study Completion 2025-05-30 (Estimated)

PRIMARY OUTCOMES:
The time to the first request of analgesia | 24 hours postoperative
  visual analogue score ≥3 by giving pethidine (50 mg IV)

SECONDARY OUTCOMES:
Total doses of analgesia | 24 hours postoperative
  (pethidine)
occurence of side effects | 24 hours postoperative
  nausea, vomiting,hypotension and bradycardia